CLINICAL TRIAL: NCT06495788
Title: Effect of High-intensity Laser Therapy on Temporalis and Masseter Muscles Activity in Patients With Myogenic Temporomandibular Joint Dysfunction
Brief Title: Effect of High-intensity Laser Therapy on Patients With Myogenic Temporomandibular Joint Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohaya Ahmed Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004882
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity laser therapy group (Experimental): Patients will receive pulsed high-intensity laser therapy in addition to conventional treatment
  Interventions: Device: High-intensity laser therapy (HILT)
- placebo high-intensity laser therapy group (Placebo Comparator): Patients will receive placebo high-intensity laser therapy in addition to conventional treatment
  Interventions: Device: placebo high-intensity laser therapy

INTERVENTIONS:
Device: High-intensity laser therapy (HILT) — * Pulsed high-intensity laser therapy (HILT) will be applied 3 sessions per week for 8 weeks with pulsed emission (1064 nm), very high peak power (3 kW), a short duration (120-150 ms), and low frequency (10-40 Hz).The probe is fixed vertically at 90° to the most painful points while the patients sit on a chair and wear safety eyewear.
  * Conventional treatment ( 3 days per week for 8 weeks).: in the form of
  * Hot pad: It will be used over the temporomandibular joint (TMJ) for 5 minutes at the beginning of each session.
  * Ultrasound therapy (US): it will be applied over the TMJ with pulsed intensity of 1.0 W/cm2 at a 1MHz frequency for 5 min/session.
  * TENS: one electrode is placed over the TMJ and the other just above the mandibular angle. it will be applied with a low frequency of 50 HZ, tolerable intensity for 15 minutes.
  * Exercise therapy: anterior, medial and lateral glide of the mandible. Each glide will be done 10-15 repetitions, 5-6 times in a session, 10 minutes as a total.
  Arms: High-intensity laser therapy group
Device: placebo high-intensity laser therapy — The same treatment procedure will be applied in the placebo group as in the experimental group, but the laser device is turned off during applications, in addition to the conventional treatment in the form of hot pad, US, TENS, and exercise therapy.
  Arms: placebo high-intensity laser therapy group

SUMMARY:
This study will be conducted to investigate the effect of high-intensity laser therapy on the temporalis and masseter muscles activity in patients with myogenic temporomandibular joint dysfunction.

DETAILED DESCRIPTION:
Temporomandibular joint dysfunction (TMD) is one of the problems that affect the quality of lifestyle through the presence of pain around the joint radiated in the face, neck, or shoulders muscles and a decrease in function of the temporomandibular joint that leads to difficulty in mastication, swallowing, earaches, dizziness, and hearing problems may sometimes be associated with TMD.

High-intensity laser therapy (HILT) is a laser with a wavelength of 1064 nm and has recently been used in the treatment of musculoskeletal diseases. Its primary effect is the analgesic effect and reactive vasodilation by affecting the cutaneous nerve endings. Another mechanism of action is based on tissue stimulation. This stimulation occurs at the level of cells, vascular tissue, interstitial tissue, and the immune system. It increases regeneration and beta-endorphin release by inducing protein synthesis in synovial fluid, thus exerting analgesic and anti-inflammatory effects.

Since there is a lack of literature studying the effect of HILT on masseter and temporalis muscles activity in patients with myogenic TMD so, this study may provide a baseline for a new technique in rehabilitation intervention in patients with myogenic TMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both gender with unilateral myogenic temporomandibular dysfunction (TMD) with trismus diagnosed and referred from maxillofacial specialist.
* Aged between 20 to 45 years old .
* Visual analogue scale (VAS) score >3 for unilateral myogenic pain of the temporomandibular joint (TMJ).
* Pain lasting at least 3 months.
* Patients were diagnosed as unilateral myogenic pain.

Exclusion Criteria:

* Previous TMJ surgery.
* History of jaw dislocation.
* History of jaw fracture.
* Previous therapy with occlusal splint.
* Concomitant therapy of bruxism.
* Presence of removable oral prosthesis.
* Metal implants in the skull.
* Presence of hearing aids.
* Malignancy.
* Pregnancy.
* Diabetic patients.
* Hypertensive patients.
* Systemic rheumatologic disease
* Systemic infection.
* Inserted cardiac pacemaker.
* Presence of coagulation disorders.
* Trigeminal neuritis.
* Cognitive dysfunction.
* Bilateral TMD.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-12 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Temporalis and masseter muscles activity | within 8 weeks
  The surface electromyography device (sEMG) (MyoTrac Infiniti 2 Channel sEMG w/Rehab Suite & Continence Suite-T9855; Quebec, Canada) at 60 Hz and Infiniti software will be used to record masseter and temporalis activity before and after the treatment program.
  patients will be instructed to clench to help the researcher to find the appropriate muscle location by their prominence. Pregelled and self-adhesive electrodes with 3 surface leads (2 recording, 1 reference) will be used. The electrode is placed over the anterosuperior to the angle of the mandible on both sides for recording masseter muscle, while for temporalis muscle, electrodes are placed above a line drawn from upper earline to canthus of the eye with interelectrode distance which is 8mm.
  sEMG Signal Analysis: Mean, median frequency, SD, root mean square, minimum, maximum, and range of muscle activity (μV) will be calculated.
Pain intensity | within 8 weeks
  Visual analogue scale (VAS), a valid and reliable measure of pain intensity will be used to measure pain intensity for all participants in both groups before and after treatment. All participants will be asked to mark their pain level on a 10-cm line that corresponds to their pain intensity on the line between "0", representing "no pain", and "10", representing "the worst pain.
Range of mouth opening | within 8 weeks
  Flexible millimeter ruler will be used to measure mouth opening for all participants in both groups before and after the treatment. Mouth opening will be evaluated by asking the patient to open their mouth as wide as possible and measuring the distance between the edges of the frontal incisors with a ruler at the incisal edge of the maxillary central incisor that is the most vertically oriented and measured vertically to the labio-incisal edge of the opposing mandibular incisor to assess the pre-post therapy maximum mouth opening (MMO). Studies reported range has been as wide as 32-62 mm (for both sexes)

SECONDARY OUTCOMES:
Limitation of Daily Function Temporomandibular Dysfunction questionnaire (LDF-TMDQ) | within 8 weeks
  Arabic version of LDF-TMDQ will be used to assess the limitation of daily function in patients with temporomandibular dysfunction in both groups before and after the treatment program. It consists of 10 items. For each item, the subject chose any one of five levels on a numerical rating scale from no problem at all (0) to extremely difficult (4 points). The total score of the 10 items, ranging from 0-40 points, will be analyzed. Internal consistency of the total scores appeared to be good at 0.78 for the 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Saleh, professor, Study Chair — Cairo University; Naglaa Awais, PHD, Study Director — Cairo University; Hala Hazzaa, professor, Study Director — Al-Azhar University; Yasser Lasheen, PHD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol